CLINICAL TRIAL: NCT03921775
Title: A Multicenter, Randomized, Single-blind, Parallel and Control Phase III Trial Evaluating the Efficacy and Safety of Remimazolam Tosilate Compared to Propofol for General Anesthesia During Elective Surgery.
Brief Title: A Clinical Study of Remimazolam Tosilate Compared to Propofol for General Anesthesia During Elective Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-RMZL-Ⅲ-GA
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia for Elective Surgery Patients
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): IV pumping of remimazolam tosilate at 6mg/kg/h for anesthesia induction and 1mg/kg/h for anesthesia maintenance
  Interventions: Drug: Remimazolam Tosilate
- Treatment B (Active Comparator): IV pumping of propofol at 120~150mg/kg/h for anesthesia induction and 3~12mg/kg/h for anesthesia maintenance
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Tosilate — For induction and maintenance of general anesthesia
  Arms: Treatment group A
Drug: Propofol — For induction and maintenance of general anesthesia
  Arms: Treatment B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of remimazolam tosilate compared to propofol for general anesthesia during elective surgery.

ELIGIBILITY:
Inclution Criteria:

1. 18~60 years, female or male
2. Patients scheduled for an elective surgical procedure(mechanical ventilation via endotracheal tube)
3. BMI: 18~30 kg/m2
4. Patients understand clearly and participate in the study voluntarily, and sign the informed consent

Exclusion criteria:

1. Patients scheduled for emergency surgery
2. Patients with a history of drug abuse and / or alcohol abuse 2 years prior to the screening period
3. One or more of the laboratory findings fall out of the limitations for this study(platelet,hemoglobin,aspartate aminotransferase,etc.)
4. Pregnant women or those in lactation period
5. Allergic to drugs used in the study
6. Patients with respiratory management difficulties (Modified Mallampati grade IV)
7. Patients have participated in other clinical trial within the 3 months prior to randomization
8. Any patient judged by the Principal Investigator (PI) or Sub-Investigator to be inappropriate for the subject for any other reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage(%) of paticipants who experienced successful anesthesia during operation in each group | Average of 2 hours

SECONDARY OUTCOMES:
Time from start of investigational medicinal product administration to loss of consciousness | Average of 2 hours
Time from stop of investigational medicinal product to MOAA/S Score=5 | Average of 2 hours
Time from stop of investigational medicinal product to Aldrete Score>9 | Average of 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China